CLINICAL TRIAL: NCT05332145
Title: Development and Proof-of-Concept Trial of a Meaning- and Theory-based Physical Activity Intervention
Brief Title: MAP to Health Pilot Study: A Physical Activity Intervention for Midlife Adults
Acronym: MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A20-287; R21AG070161 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-18 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-06

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: In Phase 1, the investigators will develop the MAP to Health web-based interview that will be used to explore what is particularly meaningful to participants, how physical activity is consistent with those goals, and what activities patients plan to engage in. Participants (N=12) will complete the interview and rate the ease of use, usefulness, intention to use, and theoretical fidelity of the intervention.
  In Phase 2, the investigators will conduct a proof-of-concept pilot trial using a double-pretest single group design. Participants (N=35) will complete a 4-week pretest monitoring period and an 8-week pilot trial of the intervention, with assessments of Self-Determination Theory mechanisms and meaning salience at pretest (-4 weeks), baseline (0 weeks), midpoint (4 weeks) and posttest (8 weeks). In addition, participants will wear accelerometers to assess physical activity during the 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention development and testing (Experimental): Phase 1 participants (N=12) will complete the MAP to Health online interview and rate the ease of use, usefulness, intention to use, and theoretical fidelity of the intervention.
  Phase 2 participants (N=35) will participate in a proof-of-concept pilot trial via a double-pretest single group design. Participants will complete a 4-week pretest monitoring period and an 8-week pilot trial of the intervention, with assessments of Self-Determination Theory mechanisms and meaning salience at pretest (-4 weeks), baseline (0 weeks), midpoint (4 weeks) and posttest (8 weeks). In addition, participants will wear accelerometers to assess physical activity during the 12 week period.
  Interventions: Behavioral: MAP to Health

INTERVENTIONS:
Behavioral: MAP to Health — In Phase 1, participants will complete the web-based interview and Aim 1 measures, assessing acceptability and usability of the intervention. The investigators will review whether the intervention appropriately gathers information needed to program theory-based, personalized text messages. After completing the measures, a list of text messages for that participant will be generated and sent to the participant for review. Participants will review the text messages and rate the extent to which the messages are personalized. In Phase 2, the investigators will conduct a proof-of-concept pilot trial in which participants will complete a 4-week pretest monitoring period and an 8-week pilot trial of the intervention, with assessments of Self-Determination Theory mechanisms and meaning salience at pretest (-4 weeks), baseline (0 weeks), midpoint (4 weeks) and posttest (8 weeks). In addition, participants will wear accelerometers to assess physical activity during the 12 weeks.

SUMMARY:
The study has two aims: (1) to develop and examine the acceptability of the technological and theoretical frameworks of MAP to Health and (2) to determine whether MAP to Health is related to changes in theoretically identified mechanisms of behavior change (meaning salience, basic psychological needs satisfaction, and internal motivation). In an exploratory aim, the study will assess how the intervention and mechanisms of change are related to changes in physical activity. Participants will be adults in midlife (ages 40-64) who are insufficiently active, are interested in increasing physical activity, do not have contraindications to engaging in physical activity, and are patients in a large healthcare system in the Midwest.

ELIGIBILITY:
Inclusion Criteria:

* Midlife (ages 40-64 at enrollment)
* Able to read and understand English
* Insufficiently active (engaging in ≥10 and ≤90 min of physical activity/week)
* Intention to increase physical activity in the next 30 days
* Has consistent access to a phone with text-messaging capability

Exclusion Criteria:

* Greater than minimal risk to starting a physical activity program (Physical Activity Readiness Questionnaire score > 0)
* Body Mass Index (BMI)≥ 40
* Currently pregnant
* Has opted out of research
* Diagnosis of metastatic cancer or cardiovascular disease
* Residing in a nursing home or long-term care facility
* Cognitive or psychiatric conditions that preclude completion of questionnaires, including dementia diagnosis
* Diagnosis of severe psychiatric disorder (e.g., Bipolar Disorder, Schizophrenia)
* Diagnosis of substance use disorder or AUDIT-C62 >3 for women or >4 for men

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Hooker, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Institute, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
If approved by HealthPartners Office for Compliance and Integrity and the HealthPartners Institutional Review Board, the investigators will also follow our local standard operating procedures for data de-identification at the conclusion of the study and provide de-identified datasets to National Institute on Aging and posted on a generalist data repository (e.g., Open Science Framework) in a preferred format. Datasets will also be provided to other qualified researchers at written request.
Supporting Information: Study Protocol, SAP, Analytic Code

RESULTS

PARTICIPANT FLOW:
Groups:
- MAP to Health Intervention: Phase 2: Phase 2 participants (N=35) will participate in a proof-of-concept pilot trial via a double-pretest single group design. Participants will complete a 4-week pretest monitoring period and an 8-week pilot trial of the intervention, with assessments of Self-Determination Theory mechanisms and meaning salience at pretest (-4 weeks), baseline (0 weeks), midpoint (4 weeks) and posttest (8 weeks). In addition, participants will wear accelerometers to assess physical activity during the 12 week period.
Period: Overall Study
Arm/Group | MAP to Health Intervention: Phase 2
Started | 35
Completed | 33
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention Testing: Participants will complete a 4-week pretest monitoring period and an 8-week pilot trial of the intervention, with assessments of Self-Determination Theory mechanisms and meaning salience at pretest (-4 weeks), baseline (0 weeks), midpoint (4 weeks) and posttest (8 weeks). In addition, participants will wear accelerometers to assess physical activity during the 12 week period.
Arm/Group | Intervention Testing
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Basic Psychological Needs Satisfaction [Mean (Standard Deviation); unit: score on a scale] — The Psychological Needs Satisfaction in Exercise Scale is a self-report measure used to assess participants' satisfaction of three basic psychological needs (autonomy, competence, and relatedness) in exercise. The scale has 18 items that participants rate on a 6-point Likert-type scale ranging from 1 (false) to 6 (true). A higher score indicates a greater sense of needs satisfaction, a better outcome. Items are averaged within and across the subscales for total scores. Population: This study used a double baseline pilot trial design. Participants completed a pre-test assessment (-4 weeks) at which time demographics were gathered for N=35 participants, defining the overall population. Four weeks later, participants completed a baseline assessment (time 0) which included N=34 participants, the start of the intervention.
  score on a scale
    Competence: number analyzed (Participants) | 34
    Competence | 4.3 (1.27)
    Autonomy: number analyzed (Participants) | 34
    Autonomy | 5.2 (0.77)
    Relatedness: number analyzed (Participants) | 34
    Relatedness | 3.7 (1.49)
Meaning Salience [Mean (Standard Deviation); unit: score on a scale] — The Meaning Awareness Scale is a 6-item self-report measure that assesses meaning salience. Participants rate the extent to which they were aware of meaning over the past day (e.g, "I was aware of the meaning in my life" on a 7-point Likert type scale ranging from 1 (rarely) to 7 (very often). Participants complete the scale on three random days during each of the four assessment periods and total scores are averaged across those three days. A higher score signifies greater meaning salience, a better outcome. Population: This study used a double baseline pilot trial design. Participants completed a pre-test assessment (-4 weeks) at which time demographics were gathered for N=35 participants, defining the overall population. Four weeks later, participants completed a baseline assessment (time 0) which included N=34 participants, the start of the intervention.
  score on a scale
    number analyzed (Participants) | 34
    (all) | 5.09 (1.48)
Autonomous Motivation [Mean (Standard Deviation); unit: score on a scale] — Autonomous motivation was measured using the Behavioral Regulations in Exercise Questionnaire, version 4. Three subscales (intrinsic, integrated, and identified) with 4 items each assess autonomous motivations for exercise on the self-determination theory continuum. Items are summed within each subscale (range, 4-28) and then subscale scores are averaged for an autonomous motivation scale, (range 4-28). Higher scores on the autonomous subscale indicate greater internalized motivation, a positive outcome. Population: This study used a double baseline pilot trial design. Participants completed a pre-test assessment (-4 weeks) at which time demographics were gathered for N=35 participants, defining the overall population. Four weeks later, participants completed a baseline assessment (time 0) which included N=34 participants, the start of the intervention.
  score on a scale
    number analyzed (Participants) | 34
    (all) | 19.78 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Meaning Salience
Description: The Meaning Awareness Scale is a 6-item self-report measure that assesses meaning salience. Participants rate the extent to which they were aware of meaning over the past day (e.g, "I was aware of the meaning in my life" on a 7-point Likert type scale ranging from 1 (rarely) to 7 (very often). Items are averaged for a total score (range, 1-7). Participants complete the scale on three random days during each of the four assessment periods and total scores are averaged across those three days. A higher score signifies greater meaning salience, a better outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MAP to Health Intervention: Phase 2
Number analyzed (Participants) | 33
score on a scale | 5.61 (1.22)

2. Primary Outcome: Basic Psychological Needs Satisfaction
Description: The Psychological Needs Satisfaction in Exercise Scale is a self-report measure used to assess participants' satisfaction of three basic psychological needs (autonomy, competence, and relatedness) in exercise. The scale has 18 items that participants rate on a 6-point Likert-type scale ranging from 1 (false) to 6 (true). Items are averaged within each subscale (autonomy, competence, and relatedness) with possible scores ranging from 1-6. Higher scores indicate greater satisfaction of autonomy, competence and relatedness, a better outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MAP to Health Intervention: Phase 2
Number analyzed (Participants) | 33
score on a scale
  Competence | 5.0 (0.86)
  Autonomy | 5.7 (0.6)
  Relatedness | 4.3 (1.6)

3. Primary Outcome: Autonomous Motivation
Description: • Autonomous motivation was measured using the Behavioral Regulations in Exercise Questionnaire, version 4. The 28-item self-report measure assesses motivations for exercise on the self-determination theory continuum. There are 7 subscales with 4 items each (intrinsic, integrated, identified, introjected - approach, introjected - avoidance, external, and amotivation). Items are summed within each subscale (total score range, 4-28). The subscales were combined using a bifurcation approach, where subscale scores were averaged into two subscales: autonomous (intrinsic, integrated, and identified, total score range 4-28) and controlled motivation (introjected-approach, introjected - avoidance, and external, total score range, 4-28). Higher scores on the autonomous subscale indicate greater internalized motivation, a positive outcome, whereas higher scores on the controlled subscale indicates greater external motivation, a negative outcome.
Time Frame: 12 weeks
Population: After enrollment of 35 study participants, one participant withdrew and one was lost to follow-up.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | MAP to Health Intervention: Phase 2
Number analyzed (Participants) | 33
score on a scale | 21.43 (5.06)

4. Primary Outcome: Technology Acceptance
Description: Participants answered 10 questions rating the extent to which they found the MAP to Health intervention easy to use (4 items) and useful (4-items) and their intentions to use the intervention in the future (2 items). Survey questions were based on previous research and modified for the purposes of this study. Participants rated each item on a scale from 1 (strongly disagree) to 5 (strongly agree). Items were averaged within each subscale, with possible total scores ranging from 1-5. A higher score represents greater technology acceptance, a better outcome.
Time Frame: within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MAP to Health Intervention: Phase 2
Number analyzed (Participants) | 32
score on a scale
  Usability | 4.28 (0.64)
  Ease of Use | 4.32 (0.76)
  Intent to Use | 3.77 (1.29)

ADVERSE EVENTS:
Time Frame: Study period: 12 weeks
Description: This study did not impose a physical activity plan, rather it encourage free choice of activities. As with any physical activity, there is a slight risk that participants could get injured during the study, but this trial was defined as a low risk study thus no adverse event/or serious adverse events were defined in the study protocol.
Arm/Group | MAP to Health Intervention: Phase 2
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT05332145/Prot_SAP_ICF_000.pdf